CLINICAL TRIAL: NCT02250222
Title: Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LGD-6972 in Healthy Subjects and in Subjects With Type 2 Diabetes Mellitus
Brief Title: Safety and Tolerability Study of Oral LGD-6972 for Type 2 Diabetes Mellitus
Acronym: L6972-02
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: L6972-02
Record Dates: First submitted 2014-09-19; First posted 2014-09-26 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — RVT-1502; SBE4-beta-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Part 1: LGD-6972 15 mg (Experimental): 15 mg LGD-6972 administered once daily (QD) for 14 days.
  Interventions: Drug: LGD-6972
- Part 1: Placebo (Captisol ®) (Placebo Comparator): Placebo administered once daily (QD) for 14 days.
  Interventions: Drug: Placebo (Captisol ®)
- Part 2: LGD-6972 5 mg (Experimental): 5 mg LGD-6972 administered orally QD for 14 days.
  Interventions: Drug: LGD-6972
- Part 2: LGD-6972 10 mg (Experimental): 10 mg LGD-6972 administered orally QD for 14 days.
  Interventions: Drug: LGD-6972
- Part 2: LGD-6972 15 mg (Experimental): 15 mg LGD-6972 administered orally QD for 14 days.
  Interventions: Drug: LGD-6972
- Part 2: Placebo (Captisol ®) (Placebo Comparator): Placebo administered orally QD for 14 days.
  Interventions: Drug: Placebo (Captisol ®)

INTERVENTIONS:
Drug: LGD-6972 — LGD-6972 sodium salt powder in Captisol ® (betadex [β-cyclodextrin] sulfobutylether sodium, NF)
  Other Names: LGD-6972 sodium oral solution
  Arms: Part 1: LGD-6972 15 mg; Part 2: LGD-6972 10 mg; Part 2: LGD-6972 15 mg; Part 2: LGD-6972 5 mg
Drug: Placebo (Captisol ®) — betadex [β-cyclodextrin] sulfobutylether sodium, NF
  Other Names: SBECD
  Arms: Part 1: Placebo (Captisol ®); Part 2: Placebo (Captisol ®)

SUMMARY:
Ligand Pharmaceuticals Incorporated is developing LGD-6972, a novel, orally-bioavailable addition to diet and exercise to improve glycemic control in adults with type 2 diabetes mellitus. The mechanism of action of LGD-6972 is to reduce the excess liver glucose production characteristic of type 2 diabetes mellitus that is a major contributor to hyperglycemia. This clinical trial will evaluate the safety and tolerability of escalating doses LGD-6972 administered daily over 2 weeks in both healthy subjects and subjects with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
This is to be a randomized, double-blind, placebo-controlled, sequential, multiple oral dose study conducted in normoglycemic healthy subjects (NHS) (Part 1) and subjects with type 2 diabetes mellitus (T2DM) who are treated with monotherapy metformin (a stable dose at randomization) along with diet and exercise (Part 2). Subjects with T2DM who are not on a stable dose of metformin but meet all other entry criteria may be enrolled in the study at the discretion of the Investigator, but must undergo a stabilization period of at least 12 weeks before determining eligibility for the study. In Part 1, a single group of healthy subjects will be dosed with repeated oral doses of 15 mg of LGD-6972 or placebo once daily (QD) for 14 days. In Part 2, a maximum of 3 groups of subjects with T2DM will be dosed with 3 sequential, increasing doses of LGD-6972 (5 mg, 10 mg or 15 mg) or placebo QD for 14 days.

ELIGIBILITY:
INCLUSION CRITERIA:

Part 1

1. Healthy, adult man or woman, 21 to 65 years of age. If the subject is a woman, she must be surgically sterile or naturally post-menopausal to be considered for enrollment.
2. Willing and able to provide written informed consent.
3. Not diabetic and has a fasting plasma glucose (FPG) between 70 mg/dL and 105 mg/dL, inclusive.
4. Good health with no significant concomitant pathology based on medical history, physical examination, electrocardiogram (ECG), routine laboratory tests (chemistry, hematology, lipid profile, international normalized ratio, and urinalysis), and vital signs.

Part 2

1. Healthy, adult man or woman, 21 to 65 years of age. If the subject is a woman, she must be surgically sterile or naturally post-menopausal to be considered for enrollment.
2. Willing and able to provide written informed consent.
3. Has T2DM according to American Diabetes Association criteria.
4. Currently on stable metformin therapy (unchanged dose for greater than or equal to 12 weeks prior to screening). At the discretion of the investigator, subjects who are drug naïve or whose metformin dose has not been stable for at least 12 weeks at screening, may be started on metformin or have their metformin dose stabilized. Following 12 weeks of stable metformin, they may undergo re screening including assessment of HbA1c and FPG (inclusion criteria 5 and 6).
5. Has an HbA1c level between 6.5% and 10.5% at screening. One retest is permitted.
6. Venous FPG is 125 mg/dL and 260 mg/dL at screening and either the Day -1 venous FPG or the Day 1 capillary blood glucose (CBG) is 115 mg/dL and 260 mg/dL. One retest is permitted.
7. Has a body mass index between 20 and 45 kg/m2, inclusive.

EXCLUSION CRITERIA:

Part 1

1. Has a recent history of drug and/or alcohol abuse.
2. Unwilling to comply with tobacco, nicotine, alcohol, and caffeine restrictions as specified in the protocol.
3. Unwilling to comply with restrictions on strenuous exercise as specified in the protocol.
4. Has history of clinically significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal (including pancreatitis), or metabolic disease requiring medical treatment or has any medical problems that pose an increased risk during the study or that may compromise the integrity of the study data.
5. Has liver transaminase levels (aspartate transaminase [AST] or alanine transaminase [ALT]) >10% of the upper limit of normal (ULN), or has creatine kinase (CK) levels >2 × ULN at screening or admission to clinic (Day -1).
6. Has a plasma triglyceride level >400 mg/dL. If triglyceride level is between 400 mg/dL and 500 mg/dL.
7. Has a recent history of uncontrolled high blood pressure or has systolic blood pressure <90 mmHg or >140 mmHg or diastolic blood pressure <60 mmHg or >90 mmHg at screening.
8. Is taking prescription or non-prescription drugs, vitamins, herbal, and dietary supplements, within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study drug, or is unwilling to refrain from taking any such medication until after the last protocol-specified blood sample. The use of acetaminophen, not to exceed a total daily dose of 1 g, is permitted up to 24 hours prior to admission to the investigational site and then prohibited until after the last protocol-specified blood sample. The use of stable hormone replacement medication by women, topical steroids, and stable thyroid medication is permitted.

Part 2

1. Has a history of hypoglycemic unawareness or recurrent hypoglycemia requiring assistance.
2. Has liver transaminase levels (AST or ALT) >10% × ULN, or has CK levels >1.5 × ULN at screening or admission to clinic (Day -1).
3. Has history of clinically significant cardiovascular, pulmonary, renal, endocrine (other than T2DM), hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal (including pancreatitis), or metabolic disease requiring medical treatment or has any medical problems that pose an increased risk during the study or that may compromise the integrity of the study data.
4. Has a recent history of uncontrolled high blood pressure or has systolic blood pressure <90 mmHg or >140 mmHg or diastolic blood pressure <60 mmHg or >90 mmHg at screening. One retest of blood pressure within 24 hours is permissible at the discretion of the Investigator. Therapy for hypertension (beta blockers excluded) that has been stable for at least one month prior to screening is permitted. At the Investigator's discretion, one anti-hypertensive medication (angiotensin converting enzyme inhibitor, angiotensin receptor blocker, hydrochlorothiazide, or dihydropyridine calcium-channel blocker) may be initiated, or the dosage of a current antihypertensive medication up titrated, in a subject with blood pressure slightly above the eligibility criterion at screening. After at least 4 weeks of stable blood pressure treatment, if the subject's blood pressure has decreased to within the 140/90 mmHg limit, the subject will be fully reassessed for eligibility.
5. Has received insulin for more than 6 consecutive days within 6 months prior to screening or has received insulin within 3 months prior to screening.
6. Has been treated with peroxisome proliferator-activated receptor gamma agonist, incretin therapy, amylin mimetics, or sodium-glucose linked transporter-2 inhibitor therapy within 12 weeks prior to screening; treatment with other diabetic medications (excluding metformin) within 3 weeks prior to screening.
7. Is taking concomitant medications. At least 3 months of stable therapy for thyroid replacement and hypercholesterolemia (gemfibrozil, Welchol, and cholestyramine are not permitted) and at least 4 weeks of stable hypertension medications (as described above) and low dose aspirin are permitted.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-10; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with one or more drug related adverse events or serious adverse events | At least 14 days after last dose
  Safety and tolerability of repeat (14 days for normoglycemic healthy subjects (NHS) and 14 days for type 2 diabetes mellitus (T2DM) subjects) and sequential increasing oral doses of LGD-6972 in NHS and subjects withT2DM will be compared to NHS and T2DM subjects receiving placebo.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile (area under the concentration curve (AUC) of LGD-6972 after repeat oral doses in NHS and in subjects with T2DM | 14 days
  Steady state PK profile (AUC) of LGD-6972 in NHS and in subjects with T2DM will be characterized and compared.
Change from baseline in fasting plasma glucose measured 24 hours after first dose and pre-dose Day 14 of treatment with LGD-6972 in NHS | 14 days
Change from baseline in fasting plasma glucagon measured 24 hours after first dose and pre-dose Day 14 of treatment with LGD-6972 in NHS | 14 days
Change from baseline in active and total glucagon-like-peptide (GLP-1) in fasting plasma measured 24 hours after first dose and pre-dose Day 14 of treatment with LGD-6972 in NHS | 14 days
Change from baseline in fasting plasma glucose measured 24 hours after first dose and at Day 14 of treatment with LGD-6972 in subjects with T2DM | 14 days
Change from baseline in fasting plasma glucagon measured 24 hours after first dose and at Day 14 of treatment with LGD-6972 in subjects with T2DM | 14 days
Change from baseline in fasting plasma insulin measured 24 hours after first dose and at Day 14 of treatment with LGD-6972 in subjects with T2DM | 14 days
Change from baseline in fasting plasma active and total GLP-1 measured 24 hours after first dose and at Day 14 of treatment with LGD-6972 in subjects with T2DM | 14 days
Change from baseline in 7-point weighted mean glucose during 14 days of treatment with different doses of LGD-6972 in subjects with T2DM | 14 days
Hemoglobin A1c response during 14 days of treatment with different dosages of LGD-6972 in subjects with T2DM | 14 days
PK profile (maximum concentration (Cmax) of LGD-6972 after repeat oral doses in NHS and in subjects with T2DM | 14 days
  Steady state PK profile (Cmax) of LGD-6972 in NHS and in subjects with T2DM will be characterized and compared.

OTHER OUTCOMES:
Change from baseline in fasting plasma glucose measured during an oral glucose tolerance test (OGTT) on Day 14 of treatment with LGD-6972 at 0.5, 1, 1.5, 2, 3, and 4 hours post-glucose load in one dose group of subjects with T2DM | 14 days
Change from baseline in fasting plasma glucagon measured during an OGTT on Day 14 of treatment with LGD-6972 at 0.5, 1, 1.5, 2, 3, and 4 hours post-glucose load in one dose group of subjects with T2DM | 14 days
Change from baseline in fasting plasma insulin measured during an OGTT on Day 14 of treatment with LGD-6972 at 0.5, 1, 1.5, 2, 3, and 4 hours post-glucose load in one dose group of subjects with T2DM | 14 days
Change from baseline in fasting plasma active and total GLP-1 measured during an OGTT on Day 14 of treatment with LGD-6972 at 0.5, 1, 1.5, 2, 3, and 4 hours post-glucose load in one dose group of subjects with T2DM | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Keith Marschke, Ph.D., Study Director — Ligand Pharmaceuticals
Locations (3):
- United States (3):
  - Celerion, Inc, Tempe, Arizona
  - Clinical Pharmacology of Miami, Inc, Miami, Florida
  - Medpace Clinical Pharmacology, Cincinnati, Ohio